CLINICAL TRIAL: NCT05532644
Title: Correlation of P-glycoprotein Polymorphisms With Microbial Metabolites in Patients With Alzheimer's Disease (AD) on Medication
Brief Title: Correlation of P-glycoprotein Polymorphisms With Microbial Metabolites in Patients With Alzheimer's Disease on Medication
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Magda Tsolaki, Professor, Aristotle University of Thessaloniki / Greek Alzheimer's Association and Related Disorders, Thessaloniki, Makedonia, Greece, Aristotle University Of Thessaloniki
Other Study IDs: MicroGeneAD
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease, P-gp, polymorphisms, microbiome, drugs, lipopolysaccharides, rhamnolipids
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients receiving cholinesterase inhibitors
  Interventions: Other: AD drugs
- Patients receiving memantine
  Interventions: Other: AD drugs
- Healthy people

INTERVENTIONS:
Other: AD drugs — AD drugs
  Groups: Patients receiving cholinesterase inhibitors; Patients receiving memantine

SUMMARY:
The importance of the proposed study concerns the understanding of the way in which each drug acts in each organism separately, both at the genome level and at the microbiome level. It is often observed that various treatments do not have the expected results in all patients, while, at the same time, new pathophysiological mechanisms for each disease are found. The involvement of the intestinal microbiome is one of these mechanisms and as it affects not only the progression of the disease but also the way in which drugs are metabolized (hence their action) should now be considered in every possible case. This led to the emergence of a new field of study related to personalized medicine, pharmacomicrobiomics. It includes microbiology, genomics, and pharmacology, and studies the changes that the human microbiome shows in drug exposure, action, and toxicity. However, this field is relatively new, and although there have been several reports of microbial biotransformation, there has been little in-depth research into the specificity of bacterial strains or the factors that can predict drug transformations. Therefore, this study will give the impetus for the individualized treatment, which will not only concern the genome (which is constantly evolving in recent years) but also the intestinal microbiome, which as mentioned above, is involved in many pathological conditions.

Importance of the study

Although a considerable number of studies have focused on the relationship between the microbiome and the pathogenesis of Alzheimer's Disease (AD), we have not seen any studies on the effect of drugs currently used in the treatment of AD (which are primarily cholinesterase inhibitors), such as rivastigmine, galantamine and donepezil and the NMDA (N-methyl-D-aspartate) glutamate receptor antagonist (memantine). There is also no reference to the composition and / or activity of the microbiome or to the effect of the latter on the pharmacokinetics and / or pharmacodynamics of these drugs. Also, although the human microbiome is influenced by genetic factors in the body, the effect of polymorphisms on the P-gp gene, which is involved in the pathophysiology of AD, the microbiome or its metabolites, has not been studied.

DETAILED DESCRIPTION:
Study design

In the proposed study, the patients will be divided into those receiving cholinesterase inhibitors (rivastigmine, galantamine and donepezil) and those receiving NMDA receptor antagonist therapy (memantine), based on the treatment they follow for AD. . A medical history of patients and controls, neuropsychological assessments using the respective questionnaires used in AD (which will be repeated at the end of the study-3 months) and a stool sample will be taken. Finally, a blood sample will be taken at the beginning of treatment to study P-gp ABCB1 gene polymorphisms and RLs and LPSs levels, and one at the end of the study to examinate drug levels RLs and LPSs levels in blood.

Duration:

Based on the required number of samples (patients and controls) the collection of these will last 6 months. Laboratory tests will take place in the next 12 months. Therefore, the main part of the study (sampling, laboratory analyzes) is expected to be completed in 18 months, while the stage of processing, analysis and verification of results is expected to last 6 months. The total duration of the study is expected to be 24 months.

Number of Subjects

135 subjects.

* 45 patients receiving treatment with cholinesterase inhibitors (rivastigmine, galantamine and donepezil).
* 45 patients receiving NMDA receptor antagonist (memantine).
* 45 healthy controls.

Patient Eligibility Screening Form (ESF):

An eligibility form documenting the patient's fulfillment of the entry criteria will be completed by the assessor. The following information will be included in the ESF:

* Patient identification: Initials (First initial of first name and first initial of surname), date of birth and Patient Identification Number.
* Written informed consent will be obtained from the subject. The informed consent form must be co-signed by the physician. The nature of the study and the potential risks associated with the trial will be explained to all subject candidates and their responsible informants.
* Signature and date: the ESF may be completed by an assessor but it is required that the principal investigator/study clinician sign and date the ESF to verify eligibility of the patient for inclusion.

Measured parameters:

For each patient who will participate in the study there should be a record of personal history that will include:

* Age
* Place of residence
* Eating habits (Mediterranean diet will be recommended)
* Smoking
* Medication followed in the last year
* Duration of the disease
* Other pathological conditions

Questionnaires

The neuropsychological assessment will include the following questionnaires, which are validated in Greek elderly population:

* Mini Mental Status Examination (MMSE)
* Montreal Cognitive Assessment (MoCA)
* Geriatrics Depression Scale (GDS)
* Functional or Cognitive Assessment scale (FUCAS)

Measurement methods

* The finding of P-gp ABCB1 gene polymorphisms will be performed with isolation of DNA with appropriate kits from the blood sample and will follow PCR technique with suitable primers and DNA electrophoresis or techniques real time PCR (taqman assay).
* Levels of RLs and LPs will be measured by the method ELISA and the use of corresponding antibodies.
* Drug levels in the blood will be measured by fluid high performance chromatography coupled to mass spectrometry (HPLC / MS).

ELIGIBILITY:
Patients with verified AD, which are monitored in the A' Neurological Clinic of AHEPA Hospital and the Hellenic Society of Alzheimer's Disease and Related Disorders (Alzheimer Hellas), are candidates for inclusion in the study. Patients should be in a mild or moderate stage of disease and should undergo a treatment (cholinesterase inhibitors or NMDA receptor antagonists) according to international guidelines. They will form the control team before receiving treatment, and there will be a group of healthy controls.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with verified AD receiving treatment
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Genetics | 6 months
  The primary target of this study is the correlation of the distribution of genotypes and haplotypes of ABCB1 polymorphisms of patients with AD with Rhamnolipids (RLs) and Polysaccharides (LPSs) levels, as well as with steady-state levels of the respective drugs in the blood.

SECONDARY OUTCOMES:
Microbiome | 6 months
  A secondary aim of this study is the comparison of the levels of RLs and LPSs as bacterial metabolites, in patients with AD following specific treatment with those of healthy controls and correlation with the course of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece